CLINICAL TRIAL: NCT05379582
Title: The Effect of Early Enteral Nutrition Feeding Process Assisted by Gastrointestinal Ultrasonography in Critically Ill Patients
Brief Title: The Effect of Early Enteral Nutrition Feeding Process Assisted by Gastrointestinal Ultrasonography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-050-02
Record Dates: First submitted 2022-04-28; First posted 2022-05-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Critical Illness; Acute Gastrointestinal Injury
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Implement nutrition therapy according to existing feeding procedures
- intervention group (Experimental): Implement nutrition therapy according a procedure assisted by gastrointestinal ultrasound
  Interventions: Other: Implement nutrition therapy according a procedure assisted by gastrointestinal ultrasound

INTERVENTIONS:
Other: Implement nutrition therapy according a procedure assisted by gastrointestinal ultrasound — Once the critical ill patients is stable, enteral nutrition was initiated following a procedure assisted by gastrointestinal ultrasound.
  Arms: intervention group

SUMMARY:
In critical ill patients, feeding protocol is one of the important factor which determines the successful implementation of enteral nutrition（EN）. Acute gastrointestinal injury(AGI) affects feeding tolerance, which greatly determines the successful implementation of feeding protocol. In our previously study, we found that transabdominal intestinal sonography is helpful to diagnosis AGI. Thus in this study ,we apply transabdominal gastrointestinal sonography to feeding protocol, to assess the feasibility of gastrointestinal sonography assisted enteral nutrition and its impact on critical ill patients.

DETAILED DESCRIPTION:
Patients meeting inclusion and exclusion criteria were randomly assigned to the intervention group and control group. During the first week of initiation of nutrition, enteral nutrition was conducted according to different procedures to observe the impact of different feeding procedures on clinical indicators

ELIGIBILITY:
Inclusion Criteria:

* The age is not less than 18 years
* within 24 hours after entering ICU
* Acute Physiology and Chronic Health Evaluation II (APACHE II) score > 8
* the estimated length of stay in ICU is more than 3 days
* informed consent

Exclusion Criteria:

* The normal anatomy of stomach, small intestine or the right colon was significantly changed (Gastrectomy, esophagectomy, pancreaticoduodenectomy, gastrointestinal bypass surgery, the presence of short bowel syndrome,etc.)
* Uncontrolled gastrointestinal bleeding
* Uncontrolled intestinal obstruction
* Uncontrolled mesenteric vascular disease
* Pregnancy
* breastfeeding
* Received enteral nutrition or parenteral nutrition within 24 hours prior to ICU admission
* Predict death within 48 hours after ICU admission
* Enrolled in this study before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Target-reaching rate through enteral route | Within first week
  percentage of participants who reach target calorie through enteral route

SECONDARY OUTCOMES:
The incidence of feeding intolerance | Within first week
The application of parenteral nutrition | Within first week
The application of prokinetic drugs | Within first week
The ues of vasoactive drugs | Within first week
Mechanical ventilation | Within first week
Continuous renal replacement | Within first week
The CRP level | Day0/1/3/5/7
Mortality | Day28、Day60、during hospitalization
ICU length of stay | During ICU stay
Length of hospital stay | During hospital stay
Platelet count | Day0,1,3,5,7
Total bilirubin | Day0,1,3,5,7
Serum creatinine | Day0,1,3,5,7

CONTACTS AND LOCATIONS:
Overall Officials: WenKui Yu, Professor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China